CLINICAL TRIAL: NCT01559233
Title: Clinical Study to Determine Safety and Efficacy of FPlus for Wrinkle Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Invasix (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FP1
Record Dates: First submitted 2012-03-17; First posted 2012-03-21 (Estimated); Last update posted 2012-03-21 (Estimated); Status verified 2012-03

CONDITIONS: Facial Wrinkles and Rhytides Reduction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- FPlus (Experimental)
  Interventions: Device: FPlus RF device for wrinkles and rhytide reduction

INTERVENTIONS:
Device: FPlus RF device for wrinkles and rhytide reduction — Six RF weekly treatments for face wrinkles and rhytides reduction using the FPlus device.
  Other Names: RF treatment

SUMMARY:
Patient demand for non-surgical, non-invasive, and no-downtime wrinkle and rhytides treatment procedures has grown dramatically over the past decade as new treatments and technologies have been introduced.

This study was performed in order to evaluate the efficacy and safety of the Invasix FPlus System, an innovative noninvasive system intended for wrinkles and rhytides treatment.

Subjects were treated for face wrinkles and rhytides reduction and followed for 3 months after last treatment. In order to evaluate treatment efficacy, pre and post treatment photos were introduced to three uninvolved physicians for blinded evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with mild to moderate facial wrinkles and rhytides .
* Males and females 21 - 65 years of age.
* Willingness to follow the treatment schedule, and have photographs taken.

Exclusion Criteria:

* Pacemaker or internal defibrillator, or other implanted metallic or electronic device.
* Permanent implant in the treated area such as metal plates and screws or silicon, unless deep enough in the periosteal plane.
* Avoid treatment if intra-dermal or superficial sub-dermal areas have been injected with Botox/HA/collagen/fat injections or other augmentation methods with bio-material during last 6 months.
* Current or history of skin cancer, or any other type of cancer, or pre-malignant moles.
* Severe concurrent conditions, such as cardiac disorders.
* Pregnancy or nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regime.
* Poorly controlled endocrine disorders, such as diabetes.
* Any active skin condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies, or use of anticoagulants in the last 10 days.
* Any facial surgery performed within 12 months prior to treatment.
* Facial dermabrasion, facial resurfacing, or deep chemical peeling within the last 3 months.
* Having received treatment with light, laser, RF, or other devices in the treated area within 6 months.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* Treating over tattoo or permanent makeup.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 69 (Actual)
Dates: Start 2011-02; Primary Completion 2012-02 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Lack of adverse events during treatments with the FPlus device and 3 months following last treatment. | 4.5 months

SECONDARY OUTCOMES:
Facial wrinkle reduction rate following 6 treatments with the FPlus device, as agreed 3 blinded dermatologists, based on Fitzpatrick wrinkle and elastosis scale. | 4.5 months

CONTACTS AND LOCATIONS:
Overall Officials: Robert Stephen Mulholland, Dr., Principal Investigator — Invasix
Locations (1):
- AestheticPlastic Surgery Practice, SpaMedica, Toronto, Canada